CLINICAL TRIAL: NCT04828382
Title: A Prospective Study Evaluating Maternal and Fetal Outcomes in the Era of Modulators
Brief Title: Prospective Study of Pregnancy in Women With Cystic Fibrosis
Acronym: MAYFLOWERS
Status: Active, not recruiting | Type: Observational
Sponsor: Amalia Magaret (Other)
Collaborators: University of Texas (Other); National Jewish Health (Other); Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor-Investigator, Amalia Magaret, Director of Statistical Research, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Other Study IDs: MAYFLOWERS-OB-20
Record Dates: First submitted 2021-03-22; First posted 2021-04-02 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Pregnancy Related; Cystic Fibrosis
Keywords: Pregnancy/obstetric health in women with cystic fibrosis; Pregnancy; CFTR modulators; Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the investigators aim to evaluate changes in lung function in women with cystic fibrosis (CF) during pregnancy and for 2 years after pregnancy based on exposure to highly effective cystic fibrosis transmembrane conductance regulator (CFTR) modulators.

DETAILED DESCRIPTION:
Advances in medical treatment, including the use of highly effective CFTR modulators have greatly increased life expectancy in women with CF, but the effects of pregnancy on women with CF are yet unknown. It is anticipated that over 90% of the CF population will be on CFTR modulators in the next few years. More knowledge about the effects of CFTR modulators in pregnancy is needed.

This is a prospective, multi-center, observational study to follow pregnant women with CF, conducted at 40 US sites. Women are enrolled in the first trimester of pregnancy and assessed every 3 months during pregnancy and during the first year after delivery, then every 6 months for an additional year. Changes in lung function over the course of pregnancy will be evaluated based on cumulative CFTR modulator use while pregnant while accounting for other factors that may influence changes in pulmonary function: baseline lung function, genotype, history of exacerbations, and pre-existing co-morbid conditions.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant, intending to continue pregnancy, enrolled in the Cystic Fibrosis Foundation Patient Registry (CFFPR)

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants will be recruited at Cystic Fibrosis Foundation's Therapeutics Development Network study sites. Pregnant women appearing for regular clinical care at these participating centers will be approached for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 285 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Forced expiratory volume at one second (FEV1) percent predicted after delivery and restart of modulators | 42 weeks
  Change in FEV1 percent predicted after delivery and restart of modulators relative to measures assessed prior to pregnancy
Forced expiratory volume at one second (FEV1) percent predicted after delivery | 42 weeks
  Change in FEV1 percent predicted after delivery relative to measures assessed prior to pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Raksha Jain, MD, Principal Investigator — University of Texas; Jennifer Taylor-Cousar, Principal Investigator — National Jewish
Locations (40):
- United States (40):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California San Diego, La Jolla, California
  - National Jewish Health, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Emory University, Atlanta, Georgia
  - Saint Luke's Cystic Fibrosis Center of Idaho, Boise, Idaho
  - Indiana University Medical Center, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Tulane University, New Orleans, Louisiana
  - John Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Brigham & Women's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - The Minnesota Cystic Fibrosis Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - The Cystic Fibrosis Center of Western New York, Buffalo, New York
  - Columbia University Cystic Fibrosis Program, New York, New York
  - University of Rochester Medical Center Strong Memorial, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital/University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cystic Fibrosis Program, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Intermountain Cystic Fibrosis Center, Salt Lake City, Utah
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Goralski JL, Talati AN, Hardisty EE, Vora NL. Pregnancy in People With Cystic Fibrosis Treated With Highly Effective Modulator Therapy. Obstet Gynecol. 2025 Jan 1;145(1):47-54. doi: 10.1097/AOG.0000000000005732. Epub 2024 Sep 19. PMID 39666984